CLINICAL TRIAL: NCT05046080
Title: Clinicopathologic and Ancillary Testing of Primary Clear Cell Carcinoma of the Cervix - a Rare Tumor
Brief Title: Clinicopathologic and Ancillary Testing of Primary Clear Cell Carcinoma of the Cervix
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-0989; NCI-2021-08814 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0989 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-08-25; First posted 2021-09-16 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Human Papillomavirus-Independent Cervical Adenocarcinoma, Clear Cell-Type

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (medical record review): Patients' medical records are reviewed retrospectively, and archival tumor tissue analyzed by immunohistochemistry and next generation sequencing.
  Interventions: Other: Electronic Health Record Review; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Other: Electronic Health Record Review — Medical records reviewed
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This study aims to provide a comprehensive report on clinicopathologic features, immunohistochemical/biomarker testing and molecular profile of cervical clear cell carcinoma. This study may help researchers learn more about the molecular profile of cervical clear cell carcinoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To perform a retrospective clinicopathologic study on patients diagnosed and treated for clear cell carcinoma of the cervix at M D Anderson Cancer Center (MDACC) and to delineate the immunohistochemical and molecular profile of these cases.

OUTLINE:

Patients' medical records are reviewed retrospectively, and archival tumor tissue analyzed by immunohistochemistry and next generation sequencing.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with clear cell carcinoma of the cervix at MDACC

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with clear cell carcinoma of the cervix, from January 1, 1985 to July 1, 2020
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2021-08-06 (Actual); Primary Completion 2026-09-29 (Estimated); Study Completion 2026-09-29 (Estimated)

PRIMARY OUTCOMES:
Clinicopathologic study on patients diagnosed and treated for clear cell carcinoma of the cervix | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Anasis Malpica, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org